CLINICAL TRIAL: NCT04269434
Title: Does Screening for Gonorrhea and Chlamydia Affect the Incidence of These Infections in Men Who Have Sex With Men Taking HIV Pre Exposure Prophylaxis (PrEP): a Randomized, Multicentre Controlled Trial
Brief Title: GonoScreen: Efficacy of Screening STIs in MSM
Acronym: GonoScreen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: ITM202002
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Neisseria Gonorrhoeae Infection; Chlamydia Trachomatis Infection
Keywords: screening
MeSH Terms: conditions — Gonorrhea

STUDY DESIGN:
Masking Description: The study statistician will be blinded until the statistical analysis plan (SAP) is approved
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Screening (No Intervention): In the screening arm, Ng/Ct results will be sent by the STI Laboratory to the study physicians and these participants will be treated and partner contact tracing will be done.
- No screening (Other): In the no screening arm, the STI Laboratory will only process the samples/report the results from the non-screening arm at the end of the study.
  Interventions: Other: No Screening

INTERVENTIONS:
Other: No Screening — the STI Laboratory will only process the samples/report the results from the non-screening arm at the end of the study.
  Arms: No screening

SUMMARY:
A Multicentre, controlled, randomized trial of 3 site (urethra, pharynx and rectum) sampling performed every 3 months (3x3) for Neisseria gonorrhoea (Ng)/Chlamydia trachomatis (Ct) screening (comparator) vs. no screening (intervention).

DETAILED DESCRIPTION:
This study is a multicentre, controlled, randomized trial of 3x3 Ng/Ct screening (comparator) vs. no screening (intervention). It will be performed in the PrEP cohorts situated at the Institute of Tropical Medicine (ITM), Hôpital Saint-Pierre (HSP), Liège University Hospital (CHU), University Hospital of Gent (UZG) and Erasmus Hospital (EH). All men in follow up at these five centres who report having had sex with another man in the previous year and are enrolled for PrEP follow up will be eligible to participate in the study. After signing informed consent participants will be randomized via a computer-generated schema to either 3x3 screening or no Ng/Ct screening. In both arms, participants will be followed up in an identical fashion including 3x3 screening. The only difference between the arms will be that in the screening arm, Ng/Ct results will be sent by the STI Laboratory to the study physicians and these participants will be treated and partner contact tracing will be done. The Sexually Transmitted Infection (STI) Laboratory will only process the samples/report the results from the non-screening arm at the end of the study. In both arms, all individuals with symptoms compatible with Ng or Ct will be tested and treated for these infections according to current best practice guidelines. At the end of the 12-month study period, participants whose most recent tests were positive for Ng or Ct will receive treatment for these.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide informed consent
* Men (born as males) and transwomen aged 18 or more
* Has had sex** with another man in the last 12 months
* Enrolled in Belgian PrEP program at ITM/HSP/EH/CHU/UZG with approval for TDF/FTC (Tenofovir disoproxil fumarate/Emtricitabine) reimbursement from a Belgian Medical Aid
* Willing to comply with the study procedures and to attend the clinic for the 3-monthly visits

Exclusion Criteria:

* Enrolment in another interventional trial
* Tests HIV-positive at screening
* Symptoms of proctitis or urethritis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1014 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Kenyon, MD, Principal Investigator — Institute of Tropical Medicine Antwerp
Locations (5):
- Belgium (5):
  - Institute of Tropical Medicine, Antwerp
  - CHU Saint-Pierre, Brussels
  - Hôpital Erasme, Brussels
  - UZGent, Ghent
  - CHU Liège, Liège

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vanbaelen T, Tsoumanis A, Florence E, Van Dijck C, Huis In 't Veld D, Sauvage AS, Herssens N, De Baetselier I, Rotsaert A, Verhoeven V, Henrard S, Van Herrewege Y, Van den Bossche D, Goffard JC, Padalko E, Reyniers T, Vuylsteke B, Hayette MP, Libois A, Kenyon C. Effect of screening for Neisseria gonorrhoeae and Chlamydia trachomatis on incidence of these infections in men who have sex with men and transgender women taking HIV pre-exposure prophylaxis (the Gonoscreen study): results from a randomised, multicentre, controlled trial. Lancet HIV. 2024 Apr;11(4):e233-e244. doi: 10.1016/S2352-3018(23)00299-0. Epub 2024 Feb 26. PMID 38423024

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started on 21st September 2020 and was completed on 4th June 2021. Participants were recruited at 5 sites (Institute of Tropical Medicine Antwerp, University Hospital Ghent, University Hospital Erasme Brussels, University Hospital Saint-Pierre Brussels and University Hospital Liège.
Period: Overall Study
Arm/Group | Screening | No Screening
Started (First Participant First Visit (FPFV)) | 506 | 508
Completed (Last Participant Last Visit (LPLV)) | 439 | 440
Not Completed | 67 | 68

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Screening | No Screening | Total
Number analyzed (Participants) | 506 | 508 | 1014
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 39 [33 to 47] | 39 [32.5 to 48] | 39 [33 to 47]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Male | 506 | 505 | 1011
  Sex: Transwoman | 0 | 3 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Number of sex partners (last 3 months) [Median (Inter-Quartile Range); unit: Number of sex partners] | 4 [2 to 8] | 4 [2 to 8] | 4 [2 to 8]
Number of sex partners (mean) [Mean (Full Range); unit: Number of sex partners] | 6.28 [0 to 100] | 7.26 [0 to 150] | 6.77 [0 to 150]
Number of unprotected sex partners in the last 3 months [Median (Inter-Quartile Range); unit: Number of unprotected sex partners] | 2 [1 to 5] | 2 [1 to 5] | 2 [1 to 5]
Number of unprotected sex partners (mean) [Mean (Full Range); unit: Number of unprotected sex partners] | 3.80 [0 to 40] | 4.28 [0 to 100] | 4.04 [0 to 100]
STI symptoms [Count of Participants; unit: Participants]
  Missing | 0 | 1 | 1
  No | 504 | 503 | 1007
  Yes | 2 | 4 | 6
Antibiotics in the last 6 months [Count of Participants; unit: Participants]
  Any | 192 | 173 | 365
  Cephalosporins | 67 | 77 | 144
  Macroloides | 81 | 94 | 175
  Penicillins | 63 | 47 | 110
  Quinolones | 11 | 5 | 16
  Tetracyclines | 57 | 54 | 111
  Other | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Ng Plus Ct Detected at Any Site Whilst Individuals Are Screened vs. Not Screened
Description: number of diagnoses of Ng plus Ct in 12 months in screening/non-screening arms divided by number of scheduled study visits with available results for the diagnosis of Ng/Ct. The denominator does not include unscheduled visits.
Time Frame: 12 months
Population: Per protocol analysis
Measure: Number (95% Confidence Interval); unit: Ng or CT cases per study visit
Arm/Group | Screening | No Screening
Number analyzed (Participants) | 357 | 344
Ng or CT cases per study visit | 0.155 [0.128 to 0.186] | 0.205 [0.171 to 0.246]
Statistical Analysis 1: Comparison: No Screening; Compared to screening group; Test type: Non-Inferiority — The "No Screening Arm" is considered non-inferior if the upper limit of the 95% Confidence Interval is less than 1.25; Incidence rate ratio = 1.318, 95% CI 2-sided [1.068 to 1.627]

2. Secondary Outcome: Cumulative Antimicrobial Exposure (Ceftriaxone/Azithromycin/Doxycycline)
Description: Number of standard doses per 1000 person-years for azithromycin, ceftriaxone and doxycycline
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: doses per 1000 person-years
Arm/Group | Screening | No Screening
Number analyzed (Participants) | 357 | 344
doses per 1000 person-years
  Azithromycin | 0.0059 [0.0055 to 0.0063] | 0.0046 [0.0043 to 0.0050]
  Ceftriaxone | 0.0008 [0.0007 to 0.0009] | 0.0004 [0.0004 to 0.0006]
  Doxycycline | 0.0081 [0.0075 to 0.0086] | 0.0044 [0.0041 to 0.0048]
Statistical Analysis 1: Comparison: No Screening; For Azithromycin. Compared to screening group; Test type: Non-Inferiority — No prespecified margin; Incidence rate ratio = 0.788, 95% CI 2-sided [0.719 to 0.863]
Statistical Analysis 2: Comparison: No Screening; For Ceftriaxone. Compared to screening group; Test type: Non-Inferiority — No prespecified margin; Incidence rate ratio = 0.561, 95% CI 2-sided [0.426 to 0.739]
Statistical Analysis 3: Comparison: No Screening; For Doxycycline. Compared to screening group; Test type: Non-Inferiority — No prespecified margin; Incidence rate ratio = 0.55, 95% CI 2-sided [0.515 to 0.588]

3. Secondary Outcome: Incidence Rate of Symptomatic Ng Plus Ct
Description: Number of diagnoses of symptomatic Ng and Ct infections over 12 months divided by number of visits
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Symptomatic infections per study visit
Arm/Group | Screening | No Screening
Number analyzed (Participants) | 357 | 344
Symptomatic infections per study visit | 0.034 [0.023 to 0.049] | 0.046 [0.032 to 0.067]
Statistical Analysis 1: Comparison: No Screening; Compared to screening group; Test type: Non-Inferiority — No prespecified margin; Incidence rate ratio = 1.373, 95% CI 2-sided [0.963 to 1.956]

4. Secondary Outcome: Incidence Rate of Syphilis
Description: Number of diagnoses of syphilis over 12 months divided by number of visits
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Syphilis cases per study visit
Arm/Group | Screening | No Screening
Number analyzed (Participants) | 357 | 344
Syphilis cases per study visit | 0.018 [0.011 to 0.029] | 0.026 [0.016 to 0.042]
Statistical Analysis 1: Comparison: No Screening; Compared to screening group; Test type: Non-Inferiority — No prespecified margin; Incidence rate ratio = 1.471, 95% CI 2-sided [0.943 to 2.299]

ADVERSE EVENTS:
Time Frame: No adverse event data collected in this study.
Description: Serious and other [non-serious] adverse events were not collected or assessed as part of the study
Arm/Group | Screening | No Screening
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT04269434/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT04269434/SAP_001.pdf